CLINICAL TRIAL: NCT07240987
Title: A Randomized Controlled Study of Mesenchymal Stem Cells in the Treatment of Chronic Kidney Diseases
Brief Title: Mesenchymal Stem Cells for Chronic Kidney Diseases
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Air Force Medicial University (Other)
Responsible Party: Principal Investigator, Li Jipeng, Principal Investigator, The First Affiliated Hospital of Air Force Medicial University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20242307
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Kidney Disease, Chronic; Diabetic Kidney Disease (DKD); Hypertensive Nephropathy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies; Hypertensive Nephropathy | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DKD (Experimental)
  Interventions: Drug: MSCs
- HN (Experimental)
  Interventions: Drug: MSCs
- non-DKD (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride
- non-HN (Placebo Comparator)
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: 0.9% sodium chloride — The control group will receive a placebo, which is an intravenous infusion of 250 mL of 0.9% sodium chloride injection.
  Arms: non-DKD; non-HN
Drug: MSCs — The experimental group will receive an intravenous injection of allogeneic MSCs at a dose of 1.0×10⁶ cells per kilogram, reconstituted with 250 mL of sodium chloride injection.
  Arms: DKD; HN

SUMMARY:
This study will evaluate the effect of intravenous injection of umbilical cord tissue derived mesenchymal stem cells (UMSCs) on the improvement of renal function in patients with chronic kidney disease (CKD) at stage 3 or 4, with the change of estimated glomerular filtration rate (eGFR) as the primary endpoint, and other changes in renal function laboratory indicators, changes in other organ system function laboratory indicators, and adverse reaction events as secondary endpoints. This trial aims to further evaluate the efficacy and safety of UMCSs in CKD patients, and provide new insights into expanding the clinical treatment strategies, delaying the progression and improving the prognosis of CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in the trial and provision of signed written informed consent
* Pathological diagnosis of diabetic nephropathy or hypertensive renal damage
* 15 ≤ eGFR < 60 mL/min/1.73m², UACR > 300 mg/g
* Age ≥ 18 years

Exclusion Criteria:

* Extremely severe anemia (hemoglobin < 30 g/L)
* Received blood product transfusion therapy within 1 month
* Autosomal dominant or recessive polycystic kidney disease (ADPKD)
* History of kidney transplant or other solid organ transplant
* Active systemic or localized infection (e.g., pneumonia, osteomyelitis)
* Allergy to stem cells themselves or stem cell-related culture medium
* History of allergic reaction to cell products (e.g., blood transfusion, platelets)
* History of coagulation disorders (thromboembolism, pulmonary embolism, deep vein thrombosis)
* History of malignancy or current malignant disease
* Elevated tumor markers (AFP, CEA, CA199, CA125, etc.)
* Pregnant women or women with plans for pregnancy within 3 months after MSC therapy
* Participation in drug-related clinical trials within the past 2 months
* Any form of drug abuse, mental illness, or other conditions considered by the investigator as potentially affecting the trial's validity or the subject's health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | From enrollment to the end of treatment at 12 months
  Efficacy Endpoints: Changes in eGFR, 24-hour urine protein, and UACR at 1, 3, 6, and 12 months will serve as primary endpoints to assess renal function improvement. Changes in other renal function parameters (e.g., quantitative urine protein, urine red blood cells, serum creatinine, cystatin C),and changes in other organ system function parameters (e.g., ECG/echocardiography, complete blood count, liver function, NT-proBNP, parathyroid hormone, 25-dihydroxyvitamin D, lymphocyte subsets) at 1, 3, 6, and 12 months will serve as secondary endpoints.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT07240987/Prot_SAP_001.pdf
  • Study Protocol: English Translation Version2 (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT07240987/Prot_002.pdf